CLINICAL TRIAL: NCT01012765
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter, 3-period Crossover Study to Compare the Effect of Indacaterol (150μg o.d.) on Inspiratory Capacity to Placebo in Patients With Moderate COPD, Using Open Label Tiotropium (18μg o.d.) as Active Control
Brief Title: Effect of Indacaterol on Inspiratory Capacity (IC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149BDE01; EUDRACT No.: 2009-013686-26 (Other: EUDRACT)
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; indacaterol; QAB149; inspiratory capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Indacaterol - placebo - tiotropium (Experimental): In treatment period 1, patients received indacaterol 150µg once daily; in treatment period 2, patients received placebo to indacaterol once daily; in treatment period 3, patients received tiotropium 18µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Placebo - Tiotropium - Indacaterol (Experimental): In treatment period 1, patients received placebo to indacaterol once daily; in treatment period 2, patients received tiotropium 18µg once daily; in treatment period 3, patients received indacaterol 150µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Tiotropium - indacaterol - placebo (Experimental): In treatment period 1, patients received tiotropium 18µg once daily; in treatment period 2, patients received indacaterol 150µg once daily; in treatment period 3, patients received placebo to indacaterol once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Placebo - indacaterol - tiotropium (Experimental): In treatment period 1, patients received placebo to indacaterol once daily; in treatment period 2, patients received indacaterol 150µg once daily; in treatment period 3, patients received tiotropium 18µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Indacaterol - tiotropium - placebo (Experimental): In treatment period 1, patients received indacaterol 150µg once daily; in treatment period 2, patients received tiotropium 18µg once daily; in treatment period 3, patients received placebo to indacaterol once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Tiotropium - placebo - indacaterol (Experimental): In treatment period 1, patients received tiotropium 18µg once daily; in treatment period 2, patients received placebo to indacaterol once daily; in treatment period 3, patients received indacaterol 150µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150µg once daily (o.d.) delivered via single-dose dry powder inhaler (SDDPI)
Drug: Tiotropium — Tiotropium 18µg o.d. delivered via a proprietary inhalation device.
Drug: Placebo — Placebo to indacaterol o.d. delivered via SDDPI

SUMMARY:
This study is being conducted to assess the effect of indacaterol (150 μg o.d.) on inspiratory capacity (IC), using placebo and open label tiotropium (18 μg o.d.) as comparators in patients with moderate chronic obstructive pulmonary disease (COPD). In particular, spirometric timepoints are included to elucidate the peak-IC in a period of approximately 4 hour post inhalation

ELIGIBILITY:
Inclusion Criteria:

* Co-operative outpatients with a diagnosis of COPD (moderate as classified by the GOLD Guidelines, 2008) and including:

  * Smoking history of at least 10 pack years
  * Post-bronchodilator FEV1 <80% and ≥50% of the predicted normal value (Visit 2).
  * Post-bronchodilator FEV1/forced vital capacity (FVC) <70% (Visit 2).

Exclusion Criteria:

* Patients who received any corticosteroid (including inhaled) for 3 months prior to screening

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Germany (21):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative site, Frankfurt am Main
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Geesthacht
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rathenow
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigator Site, Witten
  - Novartis Investigative Site, Zerbst

REFERENCES:
- [Derived] Watz H, Krippner F, Kirsten A, Magnussen H, Vogelmeier C. Indacaterol improves lung hyperinflation and physical activity in patients with moderate chronic obstructive pulmonary disease--a randomized, multicenter, double-blind, placebo-controlled study. BMC Pulm Med. 2014 Oct 4;14:158. doi: 10.1186/1471-2466-14-158. PMID 25280934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 173 participants were screened. 129 participants entered the study.
Groups:
- Tiotropium - Placebo - Indacaterol: In treatment period 1, patients received tiotropium 18µg twice daily; in treatment period 2, patients received placebo to indacaterol once daily; in treatment period 3, patients received indacaterol 150µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Indacaterol - Placebo - Tiotropium: In treatment period 1, patients received indacaterol 150µg once daily; in treatment period 2, patients received placebo to indacaterol once daily; in treatment period 3, patients received tiotropium 18µg twice daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Indacaterol - Tiotropium - Placebo: In treatment period 1, patients received indacaterol 150µg once daily; in treatment period 2, patients received tiotropium 18µg twice daily; in treatment period 3, patients received placebo to indacaterol once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Placebo - Indacaterol - Tiotropium: In treatment period 1, patients received placebo to indacaterol once daily; in treatment period 2, patients received indacaterol 150µg once daily; in treatment period 3, patients received tiotropium 18µg twice daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Placebo - Tiotropium - Indacaterol: In treatment period 1, patients received placebo to indacaterol once daily; in treatment period 2, patients received tiotropium 18µg twice daily; in treatment period 3, patients received indacaterol 150µg once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Tiotropium - Indacaterol - Placebo: In treatment period 1, patients received tiotropium 18µg twice daily; in treatment period 2, patients received indacaterol 150µg once daily; in treatment period 3, patients received placebo to indacaterol once daily. Patients received indacaterol and placebo by single-dose dry powder inhaler (SDDPI); tiotropium was delivered via a proprietary inhalation device. There was a washout period of 13 days between each period. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
Period: Treatment Period 1
Arm/Group | Tiotropium - Placebo - Indacaterol | Indacaterol - Placebo - Tiotropium | Indacaterol - Tiotropium - Placebo | Placebo - Indacaterol - Tiotropium | Placebo - Tiotropium - Indacaterol | Tiotropium - Indacaterol - Placebo
Started | 20 | 21 | 23 | 18 | 22 | 25
Completed | 17 | 21 | 21 | 15 | 19 | 25
Not Completed | 3 | 0 | 2 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Tiotropium - Placebo - Indacaterol | Indacaterol - Placebo - Tiotropium | Indacaterol - Tiotropium - Placebo | Placebo - Indacaterol - Tiotropium | Placebo - Tiotropium - Indacaterol | Tiotropium - Indacaterol - Placebo
Started | 17 | 21 | 21 | 15 | 19 | 25
Completed | 16 | 19 | 18 | 15 | 18 | 24
Not Completed | 1 | 2 | 3 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Abnormal laboratory value(s) | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 1 | 1 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Tiotropium - Placebo - Indacaterol | Indacaterol - Placebo - Tiotropium | Indacaterol - Tiotropium - Placebo | Placebo - Indacaterol - Tiotropium | Placebo - Tiotropium - Indacaterol | Tiotropium - Indacaterol - Placebo
Started | 16 | 19 | 18 | 15 | 18 | 24
Completed | 16 | 19 | 18 | 15 | 18 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Set: The safety set included all participants who received at least one dose of study medication during at least one study period.
Arm/Group | Safety Set
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Peak Inspiratory Capacity (IC) After 21 Days of Treatment
Description: IC was measured with spirometry conducted according to internationally accepted standards. Peak IC was defined as the maximum IC of the mean over the 3 values which were measured each at 30min, 2 hour, 3 hour and 4 hour post dose by body plethysmography. Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: Full analysis set (FAS) included all randomized patients who received at least one dose of study medication during at least one study period. Participants with observations after 21 days were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Indacaterol: Indacaterol 150µg once daily was administered by a single-dose dry powder inhaler (SDDPI). Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Placebo: Placebo to indacaterol was administered once daily by a single-dose dry powder inhaler (SDDPI). Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Tiotropium: Tiotropium 18µg once daily was administered via a proprietary inhalation device. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 110 | 106 | 105
Liters | 2.69 [2.64 to 2.75] | 2.48 [2.42 to 2.53] | 2.63 [2.58 to 2.69]

2. Secondary Outcome: Trough IC After 20 Days of Treatment
Description: Trough IC was measured with spirometry conducted according to internationally accepted standards. Trough IC was calculated as the mean of the three measurements of pre-dose body plethysmography (days 21, 55 and 89). Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 20 days
Population: Modified intent-to-treat (mITT) excluded patients from centers who performed invalid body plethysmography. Participants with observations after 20 days were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 87 | 83 | 84
Liters | 2.43 [2.37 to 2.50] | 2.28 [2.21 to 2.34] | 2.39 [2.32 to 2.45]

3. Secondary Outcome: Peak Residual Volume (RV) After 21 Days of Treatment
Description: Peak RV was measured with spirometry conducted according to internationally accepted standards. Peak RV was calculated as the Total Lung Capacity minus the maximum of the three Inspiratory Vital Capacity measurements which were measured each at 30 min, 2 hours, 3 hours and 4 hours post dose (at days 21, 55 and 89). Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: Modified intent-to-treat (mITT) excluded patients from centers who performed invalid body plethysmography. Participants with observations after 21 days were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 85 | 82 | 84
Liters | 3.77 [3.67 to 3.87] | 4.17 [4.07 to 4.27] | 3.79 [3.69 to 3.89]

4. Secondary Outcome: Peak Total Lung Capacity (TLC) After 21 Days of Treatment
Description: TLC was measured with spirometry conducted according to internationally accepted standards. Peak TLC was calculated as the mean of the three Functional Residual Capacity peak measurements plus the mean of the three Inspiratory Capacity measurements which were measured each at 30 min, 2 hours, 3 hours and 4 hours post dose (at days 21, 55 and 89). Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 86 | 82 | 84
Liters | 7.25 [7.16 to 7.33] | 7.38 [7.30 to 7.47] | 7.25 [7.16 to 7.33]

5. Secondary Outcome: Peak Residual Volume/Peak Total Lung Capacity (RV/TLC) Ratio After 21 Days of Treatment
Description: Peak RV/TLC ratio was measured with spirometry conducted according to internationally accepted standards. Peak RV/TLC was defined as the peak RV/peak TLC. Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 83 | 81 | 84
Ratio | 0.52 [0.51 to 0.53] | 0.57 [0.56 to 0.58] | 0.53 [0.52 to 0.53]

6. Secondary Outcome: Peak Specific Airway Resistance (sRaw) After 21 Days of Treatment
Description: Peak sRaw was measured with spirometry conducted according to internationally accepted standards. Peak sRaw was the mean of the three measurements which were measured each at 30 min, 2 hours, 3 hours and 4 hours post dose (at days 21, 55 and 89). Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa*sec
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 101 | 97 | 99
kPa*sec | 2.05 [1.89 to 2.22] | 3.08 [2.91 to 3.24] | 2.00 [1.83 to 2.16]

7. Secondary Outcome: FEV1 30 Minutes Post-dose After 21 Days of Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. FEV1 was measured 30 minutes post-dose. Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 21 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 108 | 106 | 109
Liters | 1.92 [1.89 to 1.96] | 1.68 [1.64 to 1.71] | 1.91 [1.88 to 1.95]

8. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 20 Days of Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. FEV1 was measured pre-dose after 20 days of treatment. Analysis of variance model was used with the factors: center, period, treatment, and patients within center.
Time Frame: 20 days
Population: Full analysis set (FAS) included all randomized patients who received at least one dose of study medication during at least one study period. Participants with observations after 20 days were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol | Placebo | Tiotropium
Number analyzed (Participants) | 111 | 110 | 112
Liters | 1.80 [1.77 to 1.84] | 1.61 [1.57 to 1.64] | 1.78 [1.75 to 1.82]

ADVERSE EVENTS:
Description: The safety set included all participants who received at least one dose of study medication during at least one study period.
Groups:
- Indacaterol 150ug: Indacaterol 150µg once daily was administered by a single-dose dry powder inhaler (SDDPI). Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
- Tiotropium 18ug: Tiotropium 18µg once daily was administered via a proprietary inhalation device. Use of fixed-dose combination of an anticholinergic plus a short-acting β2-agonist and use of long-acting β2-agonists were discontinued. Salbutamol rescue use was allowed during the treatment period as needed.
Arm/Group | Indacaterol 150ug | Placebo | Tiotropium 18ug
Serious Adverse Events (participants affected / at risk) | 1/118 | 1/120 | 3/119
Other Adverse Events (participants affected / at risk) | 20/118 | 16/120 | 10/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150ug (N=118) | Placebo (N=120) | Tiotropium 18ug (N=119)
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150ug (N=118) | Placebo (N=120) | Tiotropium 18ug (N=119)
NASOPHARYNGITIS (Infections and infestations) | 9 | 8 | 3
RHINITIS (Infections and infestations) | 2 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
HEADACHE (Nervous system disorders) | 2 | 3 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
HYPOTENSION (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.